CLINICAL TRIAL: NCT03667326
Title: Low-Dose Aspirin in the Postpartum Period and Endothelial Function in Patients With Preeclampsia
Brief Title: Postpartum Low-Dose Aspirin and Preeclampsia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Aleha Aziz, Assistant Professor of Obstetrics and Gynecology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AAAR9439
Record Dates: First submitted 2018-08-27; First posted 2018-09-12 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Preeclampsia Postpartum
Keywords: Aspirin
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Preeclampsia patients will be recruited and randomized to receive either Aspirin or Placebo (n = 90). Additionally, there will be healthy patients (n = 10) recruited to collect the same set of data for comparison with no intervention.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low-Dose Aspirin (LDA) Intervention Group (Active Comparator): Subjects diagnosed with severe preeclampsia prior to delivery (antepartum or intrapartum) will take 81mg of aspirin daily for up to 3 weeks postpartum, starting within 4 days after delivery.
  Interventions: Drug: Aspirin tablet
- Placebo Control Group (Placebo Comparator): Subjects diagnosed with severe preeclampsia prior to delivery (antepartum or intrapartum) will take placebo oral capsule daily for up to 3 weeks postpartum, starting within 4 days after delivery.
  Interventions: Drug: Placebo oral capsule
- Healthy Controls Group (No Intervention): Subjects who are healthy volunteers (n = 10) without severe preeclampsia prior to delivery.

INTERVENTIONS:
Drug: Aspirin tablet — Low dose aspirin, 81mg tablets, PO
  Other Names: Aspirin
  Arms: Low-Dose Aspirin (LDA) Intervention Group
Drug: Placebo oral capsule — Placebo oral capsule, PO
  Other Names: Placebo
  Arms: Placebo Control Group

SUMMARY:
The purpose of this research study is to find out whether women with severe preeclampsia taking low-dose aspirin (LDA) for 3 weeks post-delivery will experience an improvement in endothelial function (measured as flow-mediated dilation - FMD) and severity of disease, as the effects of preeclampsia can persist postpartum. Women diagnosed with severe preeclampsia prior to delivery will be enrolled and randomized to receive either low-dose aspirin (81mg) or placebo to take daily for up to 3 weeks post-delivery. Exploratory objective includes healthy control postpartum patients without preeclampsia and not on LDA during pregnancy or postpartum in comparison with the primary study population affected by preeclampsia with severe features.

DETAILED DESCRIPTION:
Preeclampsia is a serious disease of pregnancy that manifests with increased blood pressure and can affect all the organs in a woman's body. It usually develops after 20 weeks of pregnancy. There is an abnormal amount of protein in the urine and with worsening disease known as "severe features," patients can have pain in the upper abdomen, changes in vision, fluid in the lungs, an intense headache, low number of platelets in the blood, and abnormal liver or kidney function. Very high blood pressure is also considered a severe feature. The exact cause of preeclampsia is unknown but women with the condition are at increased risk for complications during pregnancy, including seizures - eclampsia. Babies are at risk of being born premature because the only cure for preeclampsia is delivery. Women who have had preeclampsia are also at increased risk of cardiovascular and kidney disease later in life, including heart attack, stroke and high blood pressure. Studies show that women at high risk for preeclampsia, i.e., have had preeclampsia in a prior pregnancy, are carrying more than one fetus, have a history of high blood pressure, kidney disease or both, have certain medical problems such as diabetes, thrombophilia or lupus, have a modestly decreased risk of disease with daily intake of low-dose aspirin starting after 12 weeks of pregnancy.

Due to the limited data available on the topic of LDA in preeclamptic patients in the postpartum period, particularly as applicable to the American population, the investigator intends to start with a small pilot study involving the collection of information on 10 women not exposed to study intervention. This will allow for confirmation of the sample size based on the baseline FMD measurements 2 days after delivery.

Investigator will also explore a small sub-study to gather information regarding baseline FMD and biomarker values for healthy control postpartum patients, unaffected by preeclampsia and not on LDA during pregnancy or postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Singleton or Multiple gestation
* Maternal age >= 18 years
* 20 0/7 weeks gestation or greater
* Severe Preeclampsia diagnosed prior to delivery

Exclusion Criteria:

* Aspirin use postpartum for other medical indication
* Lovenox, unfractionated heparin, or other anticoagulant use postpartum for an indication other than postoperative (in-house)
* Aspirin use within 7 days of planned initial FMD testing postpartum
* Hypersensitivity or allergy to Aspirin or other salicylates
* Hypersensitivity or allergy to nonsteroidal anti-inflammatory drugs (NSAIDs) - exception if taking LDA in pregnancy
* Nasal polyps
* Gastric or Duodenal ulcers, history of GI bleeding
* Severe hepatic dysfunction
* Bleeding disorders and diathesis
* Breastfeeding a newborn with low platelets (NAIT)

For sub-study patients, inclusion and exclusion criteria will be the same, with the exception of diagnosis of severe preeclampsia prior to delivery (exclusion criterion for healthy controls group).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Flow-Mediated Dilation (FMD) | Up to 3 weeks postpartum
  This is designed to measure if patients with preeclampsia with severe features diagnosed antepartum or intrapartum, will experience an increase in Flow-Mediated Dilation (FMD) - a measure of endothelial function - within 3 weeks after delivery when taking daily LDA in the postpartum period.

SECONDARY OUTCOMES:
Change in Systolic blood pressure | Within 3 weeks postpartum
  This is to measure if patients will experience a decrease in systolic blood pressure (SBP) within 3 weeks after delivery when taking daily LDA in the postpartum period.
Change in Diastolic blood pressure | Within 3 weeks postpartum
  This is to measure if patients will experience a decrease in diastolic blood pressure (DBP) within 3 weeks after delivery when taking daily LDA in the postpartum period.
Number of subjects with presentation of disease postpartum (symptoms, severe range BPs, lab abnormalities) | Up to 3 weeks postpartum
  This is to measure if patients will experience decreased severity of disease when taking daily LDA in the postpartum period.
Magnesium sulfate re-administration | Up to 3 weeks postpartum
  This is to measure if patients will experience a decreased likelihood of receiving magnesium sulfate postpartum again when taking daily LDA in the postpartum period?
Number of subjects with initiation of, increase in or addition of blood pressure medication | Up to 3 weeks postpartum
  This is to measure if patients will experience a decreased rate in initiation of/ increase in/ addition of blood pressure medication postpartum when taking daily LDA in the postpartum period.
Rate of hospital readmissions for postpartum preeclampsia | Up to 3 weeks postpartum
  This is to measure if patients will experience a decreased rate of hospital readmissions for postpartum preeclampsia when taking daily LDA in the postpartum period.

CONTACTS AND LOCATIONS:
Overall Officials: Aleha Aziz, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] The American College of Obstetricians and Gynecologists. Practice Advisory on Low-Dose Aspirin and Prevention of Preeclampsia: Updated Recommendations [Internet]. 2016. Available from: https://www.acog.org/Clinical-Guidance-and-Publications/Practice-Advisories/Practice-Advisory-Low-Dose-Aspirin-and-Prevention-of-Preeclampsia-Updated-Recommendations
- [Background] Costa AC, Reina-Couto M, Albino-Teixeira A, Sousa T. Aspirin and blood pressure: Effects when used alone or in combination with antihypertensive drugs. Rev Port Cardiol. 2017 Jul-Aug;36(7-8):551-567. doi: 10.1016/j.repc.2017.05.008. Epub 2017 Jul 3. English, Portuguese. PMID 28684123